CLINICAL TRIAL: NCT07349966
Title: A Prospective Observational Study of the Impact of Blastocyst Biopsy on Postnatal Growth in Children Born After Preimplantation Genetic Testing
Brief Title: Effects of Trophectoderm (TE) Biopsy on the Health and Development of Children Born After Preimplantation Genetic Testing (PGT) Cycles.
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Enrico Papaleo, Principal Investigator, IRCCS San Raffaele
Other Study IDs: BABYPGT
Record Dates: First submitted 2025-11-18; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Preimplantation Genetic Testing (PGT); Frozen Embryo Transfer Cycle; Assisted Reproduction Technologies; Postnatal Health
Keywords: ART; PGT; FET
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 110 children born as single live births after their mothers underwent a PGT cycle followed by frozen embryo transfer (FET).
  Interventions: Other: Questionnaire
- Controls: 220 children born as single live births after their mothers underwent only FET.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The only additional procedure involved in this study is the administration of a questionnaire to the parents, which is not part of routine clinical follow-up. The questionnaire was originally developed in the context of the Norwegian Mother and Child Cohort Study (MoBa).

SUMMARY:
This study aims to investigate the effects of trophectoderm (TE) biopsy on the health and development of children born after preimplantation genetic testing (PGT) cycles. The blastocyst biopsy is performed as part of standard clinical practice, in accordance with established protocols and current national regulations governing assisted reproduction.

ELIGIBILITY:
Inclusion Criteria for Cases:

* Child: Has completed the first year of life at the time of data collection.
* Child: Does not have any pre-existing medical conditions that significantly affect growth (weight and height).
* Mother: Able to provide informed consent for participation in the study.
* Mother: Conceived between the ages of 18 and 43.
* Mother: Achieved a singleton live birth with a single gestational sac.
* Mother: Underwent a PGT cycle followed by FET.

Inclusion Criteria for Controls:

* Child: Has completed the first year of life at the time of data collection.
* Child: Does not have any pre-existing medical conditions that significantly affect growth (weight and height).
* Mother: Able to provide informed consent for participation in the study.
* Mother: Conceived between the ages of 18 and 43.
* Mother: Achieved a singleton live birth with a single gestational sac.
* Mother: Underwent only FET.

Participants will be excluded from this study if they meet any of the following criteria:

* Mother: Unable or unwilling to sign the informed consent.
* Mother: Has undergone a fresh embryo transfer.
* Child: Missing birth weight or length/height data.

Max Age: 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will involve a total of 330 children born as single live births after their mothers underwent assisted reproduction technology (ART) treatment. The participant population includes:
  * Cases: 110 children born as single live births after their mothers underwent a PGT cycle followed by frozen embryo transfer (FET).
  * Controls: 220 children born as single live births after their mothers underwent only FET.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2028-10-27 (Estimated); Study Completion 2028-10-27 (Estimated)

PRIMARY OUTCOMES:
Impact of Blastocyst Biopsy on Postnatal Growth at One Year | 12 months of life of children
  Questionnaire

SECONDARY OUTCOMES:
Long-Term Growth After Blastocyst Biopsy | At birth of children and at 60 months of age
  Questionnaire

OTHER OUTCOMES:
Exploratory Objectives: Health and development of children at the first and fifth years of life. | At 12 and at 60 months of age
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: ENRICO PAPALEO, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Irccs San Raffaele Hospital, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alteri A, Campo G, Pagliardini L, Privitera L, Cavoretto PI, Candiani M, Papaleo E, Vigano P. The effect of vitrified-warmed blastocyst transfer on postnatal growth: a 1-year follow-up questionnaire study. Reprod Biomed Online. 2022 May;44(5):907-914. doi: 10.1016/j.rbmo.2021.12.018. Epub 2022 Jan 16. PMID 35219589
- [Background] Alteri A, Cermisoni GC, Pozzoni M, Gaeta G, Cavoretto PI, Vigano P. Obstetric, neonatal, and child health outcomes following embryo biopsy for preimplantation genetic testing. Hum Reprod Update. 2023 May 2;29(3):291-306. doi: 10.1093/humupd/dmad001. PMID 36655536
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Background] Hou W, Shi G, Ma Y, Liu Y, Lu M, Fan X, Sun Y. Impact of preimplantation genetic testing on obstetric and neonatal outcomes: a systematic review and meta-analysis. Fertil Steril. 2021 Oct;116(4):990-1000. doi: 10.1016/j.fertnstert.2021.06.040. Epub 2021 Aug 7. PMID 34373103
- [Background] Magnus P, Birke C, Vejrup K, Haugan A, Alsaker E, Daltveit AK, Handal M, Haugen M, Hoiseth G, Knudsen GP, Paltiel L, Schreuder P, Tambs K, Vold L, Stoltenberg C. Cohort Profile Update: The Norwegian Mother and Child Cohort Study (MoBa). Int J Epidemiol. 2016 Apr;45(2):382-8. doi: 10.1093/ije/dyw029. Epub 2016 Apr 10. PMID 27063603
- [Background] Ong YY, Sadananthan SA, Aris IM, Tint MT, Yuan WL, Huang JY, Chan YH, Ng S, Loy SL, Velan SS, Fortier MV, Godfrey KM, Shek L, Tan KH, Gluckman PD, Yap F, Choo JTL, Ling LH, Tan K, Chen L, Karnani N, Chong YS, Eriksson JG, Wlodek ME, Chan SY, Lee YS, Michael N. Mismatch between poor fetal growth and rapid postnatal weight gain in the first 2 years of life is associated with higher blood pressure and insulin resistance without increased adiposity in childhood: the GUSTO cohort study. Int J Epidemiol. 2020 Oct 1;49(5):1591-1603. doi: 10.1093/ije/dyaa143. PMID 32851407
- [Background] Waynforth D. Effects of Conception Using Assisted Reproductive Technologies on Infant Health and Development: An Evolutionary Perspective and Analysis Using UK Millennium Cohort Data. Yale J Biol Med. 2018 Sep 21;91(3):225-235. eCollection 2018 Sep. PMID 30258309
- [Background] Zheng W, Yang C, Yang S, Sun S, Mu M, Rao M, Zu R, Yan J, Ren B, Yang R, Guan Y. Obstetric and neonatal outcomes of pregnancies resulting from preimplantation genetic testing: a systematic review and meta-analysis. Hum Reprod Update. 2021 Oct 18;27(6):989-1012. doi: 10.1093/humupd/dmab027. PMID 34473268